CLINICAL TRIAL: NCT03925428
Title: Phase I Study of GSK525762C and Entinostat in Advanced and Refractory Solid Tumors and Lymphomas
Brief Title: Testing a New Anti-cancer Drug Combination, Entinostat and GSK525762C, for Advanced and Refractory Solid Tumors and Lymphomas
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Other - Protocol moved to Disapproved
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-02419; NCI-2019-02419 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10244 (Other: Yale University Cancer Center LAO); 10244 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2019-04-23; First posted 2019-04-24 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Ann Arbor Stage III B-Cell Non-Hodgkin Lymphoma; Ann Arbor Stage III T-Cell Non-Hodgkin Lymphoma; Ann Arbor Stage IV B-Cell Non-Hodgkin Lymphoma; Ann Arbor Stage IV T-Cell Non-Hodgkin Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Pancreatic Carcinoma; Refractory T-Cell Non-Hodgkin Lymphoma; Stage II Pancreatic Cancer AJCC v8; Stage IIA Pancreatic Cancer AJCC v8; Stage IIB Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Unresectable Pancreatic Carcinoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma; Pancreatic Neoplasms; Lymphoma, T-Cell | interventions — entinostat; molibresib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (entinostat, molibresib) (Experimental): Patients receive entinostat PO on days 1, 8, 15, and 22 and molibresib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Entinostat; Drug: Molibresib

INTERVENTIONS:
Drug: Entinostat — Given PO
  Other Names: HDAC inhibitor SNDX-275; MS 27-275; MS-275; SNDX-275
Drug: Molibresib — Given PO
  Other Names: GSK-525762A; GSK525762; I-BET 762

SUMMARY:
This phase I trial studies the side effects and best dose of GSK525762C (molibresib besylate) and entinostat in treating patients with solid tumors or lymphomas that have spread to other parts of the body (advanced) or are not responding to treatment (refractory). GSK525762C and entinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. This study may help doctors find out if giving the combination of GSK525762C and entinostat is better or worse than the usual approach for treating solid tumors or lymphomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of GSK525762C and entinostat in combination in patients with advanced and refractory solid tumors and lymphomas based on dose limiting toxicities (DLTs) of the combination of GSK525762C and entinostat.

SECONDARY OBJECTIVES:

I. To describe the safety profile of GSK525762C and entinostat in advanced and refractory solid tumors and lymphomas.

II. To determine the overall response rate (ORR) of GSK525762C and entinostat in advanced and refractory solid tumors and lymphomas.

III. To determine the progression-free survival (PFS), duration of response (DOR), and overall survival (OS) of GSK525762C and entinostat in this patient population.

EXPLORATORY OBJECTIVES:

I. To assess the effect of GSK525762C and entinostat therapy on apoptosis, as measured by an apoptosis multiplex immunoassay.

II. To assess the effect of GSK525762C and entinostat therapy on c-MYC and YAP1 as measured by ribonucleic acid (RNA) and protein expression.

III. To assess the effect of GSK525762C and entinostat therapy on tumor burden and gene expression patterns as measured by whole exome sequencing (WES) and RNA sequencing (RNASeq) on circulating tumor deoxyribonucleic acid (DNA) (ctDNA) specimens.

OUTLINE: This is a dose-escalation study.

Patients receive entinostat orally (PO) on days 1, 8, 15, and 22, and molibresib PO once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have advanced or refractory solid tumor or lymphoma (all B cell lymphomas and T cell lymphomas other than natural killer [NK]-cell lymphoma).
* For patients in the dose expansion cohort:

  * Cohort A: Patients must have locally advanced, unresectable OR metastatic pancreatic cancer refractory to standard therapy.
* Patients must have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
* Patients should have received previous therapy with at least one combination chemotherapy regimen for metastatic disease.
* Patients with lymphoma must have exhausted or refused potential curative therapy prior to enrolling.
* Weight of >= 35 kg.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 50%).
* Hemoglobin >= 9.0 g/dL (within 14 days prior to administration of study treatment).
* Absolute neutrophil count (ANC) >= 1,500/mcL (within 14 days prior to administration of study treatment).
* Platelets >= 100,000/mcL (within 14 days prior to administration of study treatment).
* Total bilirubin =< institutional upper limit of normal (ULN) (within 14 days prior to administration of study treatment).
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (within 14 days prior to administration of study treatment).
* Serum creatinine clearance > 50 mL/min (within 14 days prior to administration of study treatment).
* Serum bilirubin =< 1.5 x institutional ULN (within 14 days prior to administration of study treatment).
* Creatinine =< institutional ULN (within 14 days prior to administration of study treatment) OR
* Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73m^2 as measured by the Cockcroft-Gault equation (within 14 days prior to administration of study treatment).
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with treated brain metastases are eligible if follow-up brain imaging at least 4 weeks after central nervous system (CNS)-directed therapy shows no evidence of progression.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association functional classification. To be eligible for this trial, patients should be class 2B or better.
* Patients must be able to swallow and retain orally administered medication.
* Women of childbearing potential must have a negative pregnancy test within 7 days of starting treatment.
* The effects of entinostat and GSK525762C on the developing human fetus are unknown. For this reason and because HDAC inhibitor (HDACi) and BET inhibitor (BETi) agents are known to be teratogenic, women of child-bearing potential and their male partner must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for 7 months after completion of entinostat and GSK525762C administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of entinostat and GSK525762C administration.
* Patients must have tumors determined to be easily accessible for biopsy and must be willing to have serial biopsies. Tumor biopsies will be performed on the most accessible biopsiable site of disease. All possible precautions to avoid complications will be taken, including discussions in multidisciplinary meetings, if needed. If a biopsy cannot be performed safely (e.g. there is no safely accessible biopsiable tumor tissue) or biopsy does not yield sufficient tissue for analysis, participation is still allowed.
* Patients on both therapeutic and prophylactic anticoagulation may participate as long as they have no history of clinically significant bleeding while on anticoagulation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had any anti-cancer therapy within 14 days (or 5 half-lives, whichever is longer) prior to the first dose of the investigational products.
* Patients who have received radiation therapy within 21 days prior to the first dose of the investigational products.
* Patients who have a diagnosis of NK cell lymphoma.
* Patients who have not recovered from adverse events due to prior anti-cancer therapy. Toxicities should have recovered to =< grade 1, excluding alopecia, or should be stable chronic grade 2 toxicities that do not overlap with presumed toxicities of entinostat or GSK525762C.
* Patients who are receiving any other investigational agents.
* Patients with known untreated or symptomatic brain or leptomeningeal metastases are excluded. Patients with previously treated central nervous system (CNS) metastasis may be included provided that they have stable CNS disease for at least 4 weeks (confirmed by imaging) without symptoms and are off corticosteroids (above physiologic dose) for that indication.
* Patients with significant malabsorption or nausea and vomiting that would interfere with oral therapies.
* Patients with bleeding diathesis or clinically significant bleeding within the prior 6 months.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to entinostat (e.g. medications that have a benzamide structure [tiapride, remoxipride, clebopride] or GSK525762C [e.g. benzodiazepines]).
* Patients receiving any medications or substances that are strong inhibitors or strong inducers of CYP3A4 are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Patients with uncontrolled intercurrent illness.
* Patients with a history of clinically significant bleeding.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because entinostat is an HDACi and GSK525762C is a BETi with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with entinostat or GSK525762C, breastfeeding should be discontinued throughout the treatment period and for at least 28 days following the last dose of study treatment if the mother is treated with entinostat or GSK525762C.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | At 28 days
  Assesses with dose limiting toxicities. Descriptive statistics, including means, standard deviations, and ranges for continuous parameters, as well as percentages and frequencies for categorical parameters, will be presented.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  Graded per Common Terminology Criteria for Adverse Events version 5.0. National Cancer Institute toxicity grade 3 and grade 4 laboratory abnormalities will be listed.
Overall response rate (ORR) | Up to 2 years
  The exact two-sided 95% confidence intervals (CIs) for the RR will be reported.
Progression-free survival | Up to 2 years
  Will be estimated using the Kaplan-Meier method with the 95% CIs. The CI based on Greenwood's variance will be reported. In addition, the possible risk factors will be compared for survival with log-rank test.
Overall survival | Up to 2 years
  Will be estimated using the Kaplan-Meier method with the 95% CIs. The CI based on Greenwood's variance will be reported. In addition, the possible risk factors will be compared for survival with log-rank test.
Duration of response | Up to 2 years
  The 95% CIs for the duration of response will be reported.

OTHER OUTCOMES:
Effect of GSK525762C and entinostat combination therapy on apoptosis rate | Up to 2 years
  Measured by an apoptosis multiplex immunoassay. Statistical and bioinformatic data analysis for laboratory non-omics data and clinical data will utilize the following general strategies, as appropriate. For single time-point lab data, tests of hypotheses concerning within-group comparisons will be completed using the paired t-test or Wilcoxon signed-rank test for continuous parameters of interest, or McNemar's Chi-square test for categorical parameters of interest. Between-group comparisons will be assessed using either analysis of variance (ANOVA) with adjusted least squares means or Fisher's exact test, for continuous or categorical variables of interest, respectively. For count or binary multiple time-points or correlated data, tests of between-group comparisons will be completed using the generalized estimating equation (GEE) statistical procedure for longitudinal data analysis with multiple observable vectors for the same subject.
Effect of GSK525762C and entinostat combination therapy on c-MYC expression | Up to 2 years
  Measured by ribonucleic acid (RNA) and protein expression. Statistical and bioinformatic data analysis for laboratory non-omics data and clinical data will utilize the following general strategies, as appropriate. For single time-point lab data, tests of hypotheses concerning within-group comparisons will be completed using the paired t-test or Wilcoxon signed-rank test for continuous parameters of interest, or McNemar's Chi-square test for categorical parameters of interest. Between-group comparisons will be assessed using either ANOVA with adjusted least squares means or Fisher's exact test, for continuous or categorical variables of interest, respectively. For count or binary multiple time-points or correlated data, tests of between-group comparisons will be completed using the GEE statistical procedure for longitudinal data analysis with multiple observable vectors for the same subject.
Effect of GSK525762C and entinostat combination therapy on YAP1 expression | Up to 2 years
  Measured by RNA and protein expression. Statistical and bioinformatic data analysis for laboratory non-omics data and clinical data will utilize the following general strategies, as appropriate. For single time-point lab data, tests of hypotheses concerning within-group comparisons will be completed using the paired t-test or Wilcoxon signed-rank test for continuous parameters of interest, or McNemar's Chi-square test for categorical parameters of interest. Between-group comparisons will be assessed using either ANOVA with adjusted least squares means or Fisher's exact test, for continuous or categorical variables of interest, respectively. For count or binary multiple time-points or correlated data, tests of between-group comparisons will be completed using the GEE statistical procedure for longitudinal data analysis with multiple observable vectors for the same subject.
Effect of GSK525762C and entinostat combination therapy on tumor burden | Up to 2 years
  As measured by whole exome sequencing and RNA sequencing (RNASeq) on circulating tumor deoxyribonucleic acid (DNA) specimens.
Effect of GSK525762C and entinostat combination therapy on gene expression patterns | Up to 2 years
  As measured by whole exome sequencing and RNASeq on circulating tumor DNA specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M LoRusso, Principal Investigator — Yale University Cancer Center LAO

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm